CLINICAL TRIAL: NCT03147170
Title: Use of NT-proBNP as a Biomarker to Treat Salt Sensitive in Hypertensive Individuals
Brief Title: A Biomarker to Detect Salt Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1512M81431
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Hypertension Uncomplicated; Pre Hypertension
MeSH Terms: conditions — Prehypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: High and low salt diets — Effects of high and low salt diets on blood pressure in individuals with normal and elevated levels of NT-proBNP

SUMMARY:
The investigators are proposing that individuals with elevated levels of NT-proBNP are resistant to natriuretic peptides and are unable to handle sodium loads and maintain optimal blood pressure values.The investigators will test this hypothesis by comparing the blood pressure response to low and high salt diets in individuals with pre- or hypertension and who have normal or elevated levels of NT-proBNP. The investigators expect that blood pressure values in those with normal levels of NT-proBNP will not change with high salt diets, whereas, in those with elevated levels of NT-proBNP, blood pressure values will increase significantly when exposed to high salt diets.

DETAILED DESCRIPTION:
Natriuretic peptides (NPs) are molecules that regulate blood pressure by inducing natriuresis and vasodilation. We have shown that higher baseline levels of NT-proBNP are associated with the development of hypertension and humans elevated NT-proBNP levels demonstrate resistance to the action of NPs and are unable to handle high dietary sodium loads. These findings have led us to propose that pre-hypertensive or newly diagnose hypertensive individuals, free of overt cardiovascular disease, who have elevated levels of NT-proBNP will experience a substantial rise in total body water and arterial blood pressure when exposed to a high sodium load. If this hypothesis holds true, then NT-proBNP could be used as a biological marker to identify salt sensitivity and for the prescription of low sodium diets to hypertensive individuals.

Research design: Individuals with physiological levels of NT-proBNP (40 - 90 pg/mL) and those with elevated levels (> 120 pg/mL) will be recruited to participate in a randomized crossover feeding study designed to treat patients with hypertension. A total of 8 participants, per group, will be exposed to two 10 days-phases of either a low sodium load (LS) of 50 mmol/day or a high sodium load (HS) of 250 mmol/day in random order and compare the blood pressure response to different sodium loads between the two NT-proBNP categories. Salt sensitivity is defined as a change in mean arterial blood pressure of ≥ 10% between the low and high sodium load. At the end of each phase, participants will be tested on a variety of anthropometric, blood and urinary measurements.

Variables measured: Total body water will be determined using bioelectrical impedance from Valhalla Scientific body comp scale®. Blood pressure monitors will be provided to each participant for measurement and record their own blood pressure twice daily for the duration of the study. In addition, at the end of each of the two sodium loading phases, trained personnel will measure BP three time using standard procedures, following an 8 hour fast and a 10 minute rest period at the clinic. Laboratory measurements. Blood and urine analysis will be performed at the start and end of each salt loading phase at the Advanced Research and Diagnostic Laboratory (ARDL). NT-proBNP will be measured using the Roche-Elecsys proBNP® (Roche Diagnostics, Indianapolis, IN). This method has a range of values that extends from 1 - 25000 pg/mL and the intra-assay precision is below 4% and the CV and interassay precision below 5% 21. Plasma BNP will be measured on a Siemens Advia Centaur instrument using a chemiluminescent immunoassay which has a minimal detection limit of 1.9 pg/mL and a CV of 3.4%. cGMP will be measured using a competitive enzyme immunoassay by Bio-Techne (Minneapolis, MN) intra essay CV is 7%. NT-proBNP will be measured using the Roche-Elecsys proBNP® (Roche Diagnostics, Indianapolis, IN). This method has a range of values that extends from 1 - 25000 pg/mL and the intra-assay precision is below 4% CV and inter-assay precision below 5% 21.

Anticipated results and future studies. Individuals with elevated NT-proBNP will have a significant increase in mean blood pressure and total body water (salt sensitive individuals) and a greater BNP/cGMP ratio when compared to those with physiological levels of NT-proBNP.

Power analysis shows that for a randomized cross-over study we would need 25 individuals per group for a 90% power.

ELIGIBILITY:
Inclusion Criteria:

1. Systolic blood pressure > 120 and < 160 mmHg
2. Diastolic blood pressure > 80 and < 100 mmHg
3. Not on hypertensive medications
4. NT-proBNP between 40 - 99 pg/mL (healthy levels)
5. NT-proBNP > 120 pg/mL (elevated levels)

Exclusion Criteria:

1. Physician reported diabetes or on insulin or oral hypoglycemic agents
2. BMI > 40kg/m2
3. Age < 30 or > 75 years
4. Presence of cardiovascular disease or chronic kidney disease
5. Chronic obstructive pulmonary disease or pulmonary arterial hypertension
6. Aldosterone secreting disorder
7. Estimated energy intake greater than 3400 calories
8. Pregnancy
9. Individuals with pacemakers

Ages: 30 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Pre- or hypertensive individuals without chronic complications, between the ages of 30 and 75 years, not on blood pressure lowering medications.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | 9 weeks
  Difference in blood pressure before and after diets periods and comparison between those with normal and elevated blood levels of NT-proBNP.

SECONDARY OUTCOMES:
Ratio of BNP/cGMP | 9 weeks
  Difference in BNP/cGMP before and after diets periods and comparison between those with normal and elevated blood levels of NT-proBNP.

CONTACTS AND LOCATIONS:
Overall Officials: Otto A Sanchez, MD PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided